CLINICAL TRIAL: NCT04667728
Title: The Effects of Professional Continuous Glucose Monitoring as an Adjuvant Educational Tool in Patients With Type 2 Diabetes and Poor Glycemic Control
Brief Title: Professional Continuous Glucose Monitoring as an Adjuvant Educational Tool for Improving Glycemic Control in Patients With Type 2 Diabetes.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Seguridad y Servicios Sociales de los Trabajadores del Estado (Other Government)
Collaborators: Medtronic, PLC (Unknown)
Responsible Party: Principal Investigator, Dulce Adelaida Rivera Avila, Principal Investigator, Instituto de Seguridad y Servicios Sociales de los Trabajadores del Estado
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 318.17
Record Dates: First submitted 2020-12-08; First posted 2020-12-16 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: professional continuous glucose monitoring; educational tool; glycemic control
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Intervention Model Description: A three-month quasi-experimental study with an intervention and control group and ex-ante and ex-post evaluations
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (IGr) (Experimental): The IGr participants wore a professional continuous glucose monitoring (CGM) sensor (iPro™2) during the first six days of the study. Following this period, IGr participants had a medical consultation for the CGM results and treatment adjustments. Additionally, they received a personalized diet plan from a dietitian. After three months, the IGr participants again wore the CGM sensor for one week. These participants also followed the regular institutional Comprehensive Diabetes Care program care plan.
  Interventions: Device: Professional continuous glucose monitoring (CGM) sensor (iPro™2)
- control group (CGr) (No Intervention): The control group followed the regular institutional Comprehensive Diabetes Care program care plan.

INTERVENTIONS:
Device: Professional continuous glucose monitoring (CGM) sensor (iPro™2) — Professional continuous glucose monitoring (CGM) sensor (iPro™2) following treatment adjustments and personalized diet plan
  Arms: intervention group (IGr)

SUMMARY:
The investigators conducted a three-month quasi-experimental study with an intervention and control group and ex-ante and ex-post evaluations in one family medicine clinic in Mexico City. Participants were type 2 diabetes patients with HbA1c>8 mg/dL attending a comprehensive diabetes care program (MIDE). In addition to the program, the intervention group wore a professional CGM sensor (iPro™2) during the first six days of the study. Following this period, intervention group participants had a medical consultation for the CGM results and treatment adjustments. Additionally, the intervention group participants received an educational session and a personalized diet plan from a dietitian. After three months, the intervention group again wore the CGM sensor for one week. The primary outcome variable was HbA1c level measured at baseline and three months after the CGM intervention. The investigators analyzed the effect of the intervention on HbA1c levels by estimating the differences-in-differences treatment effect. Additionally, baseline and three-month CGM and dietary information was recorded for the intervention group and analyzed using the Student's paired t-test and mixed-effects generalized linear models to control for patients' baseline characteristics.

DETAILED DESCRIPTION:
From May to October 2017, the investigators conducted a three-month pilot study with intervention and control groups and ex-ante and ex-post evaluations in one ISSSTE family medicine clinic in Mexico City. Patients with type 2 diabetes in the comprehensive diabetes care program (MIDE) who were older than 20 years of age and had HbA1c> 8 mg/dL were considered eligible participants for the study; those who agreed to participate, were required to sign an informed consent. In May and June, the investigators invited all consecutive type 2 diabetes patients who attended the MIDE program to join the intervention group; the investigators followed the same protocol in July and August to assemble the control group.

The control group followed the MIDE care plan, consisting of at least two consultations with a medical doctor and HbA1c measurements at baseline and three months later, as well as weekly self-care educational group activities. The baseline consultation included a review of HbA1c levels and treatment adjustments.

At the beginning of the study, the intervention group had a professional CGM device (iPro™2, Medtronic, USA) inserted subcutaneously for six days. Before the CGM insertion, the intervention group received a training session on how to use and calibrate the device through three daily glucometer readings of capillary glucose. Moreover, intervention group patients were trained to record daily information on their medications, including the times and dosages taken; their diet, including the foods and portions consumed; and their physical activity practices. After six days of device use, intervention group participants had a consultation with a family physician trained in diabetes to interpret the CGM report results and adjust their treatment. In addition, a dietitian provided an educational session and personalized diet plan guided by the CGM results. Participants in the intervention group were also advised to attend regular MIDE program activities. After three months, the intervention group wore the sensor again and their HbA1C levels were measured.

After the three-month study period, the intervention and control groups continued their participation in the MIDE program. The primary outcome variable was HbA1c level measured at baseline and three months after the CGM intervention. The investigators analyzed the effect of the intervention on HbA1c levels by estimating the differences-in-differences treatment effect. Additionally, baseline and three-month CGM and dietary information was recorded for the intervention group and analyzed using the Student's paired t-test and mixed-effects generalized linear models to control for patients' baseline characteristics.

ELIGIBILITY:
Inclusion Criteria:

Patients with type 2 diabetes with HbA1c>8 mg/dL, without diagnosis of a memory disorder who agreed to participate and signed an informed consent form

Exclusion Criteria:

* None

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2017-05-30 (Actual); Primary Completion 2017-10-30 (Actual); Study Completion 2017-10-30 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in HbA1c at 3 Months | Baseline and 3 months
  Hemoglobin A1c (%)

OTHER OUTCOMES:
Change From Baseline in time in range at 3 Months | Baseline and 3 months
  Percentage of time that patients' continuous glucose monitoring (CGM) glucose readings were in the target range (70-150mg/dl)
Change From Baseline in time in hyperglycemic range at 3 Months | Baseline and 3 months
  Percentage of time the patient was in hyperglycemic range (>150 mg/dl)
Change From Baseline in time in hypoglycemic range at 3 Months | Baseline and 3 months
  Percentage of time the patient was in hypoglycemic range (<70mg/dl)
Change From Baseline in average glucose levels at 3 Months | Baseline and 3 months
  Average glucose levels (mg/dl)
Change From Baseline in glucose variability at 3 Months | Baseline and 3 months
  Glucose variability measured through standard deviation
Change From Baseline in percentage of the area over the blood concentration-time curve at 3 Months | Baseline and 3 months
  Percentage of the area over the blood concentration-time curve
Change From Baseline in percentage of the area under the blood concentration-time curve at 3 Months | Baseline and 3 months
  Percentage of the area under the blood concentration-time curve
Change From Baseline in daily total caloric intake at 3 Months | Baseline and 3 months
  Daily total caloric intake (Kcal)
Change From Baseline in daily carbohydrates intake at 3 Months | Baseline and 3 months
  Daily carbohydrates intake (Kcal)
Change From Baseline in daily proteins intake at 3 Months | Baseline and 3 months
  Daily proteins intake (Kcal)
Change From Baseline in daily fat intake at 3 Months | Baseline and 3 months
  Daily fat intake (Kcal)

CONTACTS AND LOCATIONS:
Locations (1):
- Clínica de Medicina Familiar Oriente, México, Mexico

IPD SHARING:
Plan to Share IPD: No
There is no a plan to make individual participant data (IPD) available to other researchers.

REFERENCES:
- [Background] Carlson AL, Mullen DM, Bergenstal RM. Clinical Use of Continuous Glucose Monitoring in Adults with Type 2 Diabetes. Diabetes Technol Ther. 2017 May;19(S2):S4-S11. doi: 10.1089/dia.2017.0024. PMID 28541137
- [Background] Park C, Le QA. The Effectiveness of Continuous Glucose Monitoring in Patients with Type 2 Diabetes: A Systematic Review of Literature and Meta-analysis. Diabetes Technol Ther. 2018 Sep;20(9):613-621. doi: 10.1089/dia.2018.0177. Epub 2018 Aug 10. PMID 30095980
- [Background] Taylor PJ, Thompson CH, Brinkworth GD. Effectiveness and acceptability of continuous glucose monitoring for type 2 diabetes management: A narrative review. J Diabetes Investig. 2018 Jul;9(4):713-725. doi: 10.1111/jdi.12807. Epub 2018 Mar 1. PMID 29380542
- [Background] Bruttomesso D, Laviola L, Avogaro A, Bonora E, Del Prato S, Frontoni S, Orsi E, Rabbone I, Sesti G, Purrello F; of the Italian Diabetes Society (SID). The use of real time continuous glucose monitoring or flash glucose monitoring in the management of diabetes: A consensus view of Italian diabetes experts using the Delphi method. Nutr Metab Cardiovasc Dis. 2019 May;29(5):421-431. doi: 10.1016/j.numecd.2019.01.018. Epub 2019 Feb 10. PMID 30952574
- [Derived] Rivera-Avila DA, Esquivel-Lu AI, Salazar-Lozano CR, Jones K, Doubova SV. The effects of professional continuous glucose monitoring as an adjuvant educational tool for improving glycemic control in patients with type 2 diabetes. BMC Endocr Disord. 2021 Apr 23;21(1):79. doi: 10.1186/s12902-021-00742-5. PMID 33888117